CLINICAL TRIAL: NCT03804788
Title: The Impact of Insomnia Treatment on Heavy Alcohol Use Among Returning Veterans
Brief Title: The iTAP Study for Veterans
Acronym: iTAP-V
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Mary E Miller, Professor, Psychiatry, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2014239; K23AA026895 (NIH)
Record Dates: First submitted 2019-01-09; First posted 2019-01-15 (Actual); Results first posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2024-12

CONDITIONS: Insomnia; Alcohol; Harmful Use
Keywords: alcohol; drinking; sleep; insomnia; veteran
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to receive sleep hygiene or to participate in sessions of individual Cognitive Behavioral Therapy for Insomnia (CBT-I).
Who Masked: Participant, Outcomes Assessor
Masking Description: PI Miller will be blind to participant assignment because the project manager will inform study therapists of participant assignment to conditions. PI Miller and study therapists will be blinded to assessment outcomes, and assessment RAs will be blinded to participant condition. All participants will be told that they are receiving treatment for insomnia in order to blind them to condition assignment (sleep hygiene will be described as "brief" insomnia treatment, and CBT-I will be described as the "most intense" treatment).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBT-I (Experimental): Individual Cognitive Behavioral Therapy for Insomnia (CBT-I) delivered once a week for six (6) weeks.
  Interventions: Behavioral: Cognitive Behavioral Therapy for Insomnia; Behavioral: Sleep Hygeine
- Sleep Hygiene (Active Comparator): Sleep hygiene handout delivered once to all participants.
  Interventions: Behavioral: Sleep Hygeine

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy for Insomnia — Cognitive Behavioral Therapy for Insomnia (CBT-I). Participants assigned to the CBT-I condition will attend 1-hour individual sessions of CBT-I once a week for five weeks. A sixth week of treatment will be included - and scheduled for the same date as the post-treatment assessment - if the participant and research team agree that it would be beneficial (e.g., if a participant has difficulty grasping cognitive therapy concepts). Consistent with clinical guidelines (Schutte-Rodin, Broch, Buysse, Dorsey, & Sateia, 2008), treatment will include stimulus control (e.g., limit use of bed to sleep or sexual activity, get out of bed if lying awake for more than 20 minutes), sleep restriction (limit time in bed to amount of time spent sleeping on a typical night), sleep hygiene (e.g., avoid exercise within 2 hours of bedtime, create cool and dark sleep environment), relaxation training, and cognitive restructuring.
  Other Names: (CBT-I)
  Arms: CBT-I
Behavioral: Sleep Hygeine — All participants will receive a one-page handout on sleep hygiene that includes personalized normative feedback on their alcohol use. This is the only intervention that participants assigned to the Sleep Hygiene condition will receive and is consistent with what may be expected as standard care in a doctor's visit with a primary care physician.

SUMMARY:
This project aims to evaluate improvement of insomnia as a mechanism of improvement in alcohol use outcomes.

DETAILED DESCRIPTION:
More than half of returning Veterans who screen positive for hazardous drinking report clinically significant symptoms of insomnia. In turn, insomnia symptoms have been associated with increased risk of alcohol-related problems, perhaps due to insomnia-related impairments in executive functioning, negative emotionality, and craving. The proposed project aims to examine improvements in insomnia as a mechanism for improvement in alcohol use among heavy-drinking Veterans with insomnia. Forty-four returning Veterans who report heavy drinking (≥4/5 drinks per occasion for women/men) and have insomnia based on DSM-5 and research diagnostic criteria will participate in a randomized pilot trial. Participants will be randomly assigned to receive personalized normative alcohol feedback in the context of one of two treatment conditions: CBT-I (n = 22) or a sleep hygiene education control (SH; n = 22). Outcomes will be assessed at the end of the active intervention period (6 weeks), mid-treatment (after 3 sessions), and at 3 months post-intervention. Outcomes of interest include insomnia severity, total wake time, sleep quality, drinking quantity/frequency, alcohol-related consequences, executive functioning, negative affect, emotion regulation, craving for alcohol, and use of alcohol as a sleep aid.

ELIGIBILITY:
Inclusion criteria:

* Veteran deployed for military service after September 11, 2001
* 1+ heavy drinking episode (4/5+ drinks in 2 hours for women/men) in past 30 days
* DSM-5 and research diagnostic criteria for Insomnia Disorder

Exclusion Criteria:

* Inability to provide informed consent
* Cognitive impairment
* Contraindications for CBT-I (mania or seizure disorder)
* Untreated sleep disorder requiring more than behavioral treatment for insomnia
* Engagement in overnight shift work at baseline
* Care of a child under 1 year of age
* Severe or untreated psychiatric disorder that requires immediate clinical attention
* Current behavioral treatment for insomnia or alcohol use
* Initiation of sleep medication in the past 6 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2019-04-04 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Missouri-Columbia, Columbia, Missouri, United States

REFERENCES:
- [Derived] Miller MB, Carpenter RW, Shoemaker SD, Moskal KR, Borsari B, Pedersen ER, Bartholow BD, Steinley D, McCrae CS. Cognitive behavioral therapy for insomnia among heavy-drinking veterans: a randomized pilot trial. Sleep Adv. 2025 Jun 10;6(2):zpaf037. doi: 10.1093/sleepadvances/zpaf037. eCollection 2025 Apr. PMID 40575624

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Heavy-drinking Veterans were recruited via online digital marketing between April 2019 and August 2023.
Period: Overall Study
Arm/Group | CBT-I | Sleep Hygiene
Started | 38 | 33
Completed | 38 | 33
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CBT-I | Sleep Hygiene | Total
Number analyzed (Participants) | 38 | 33 | 71
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.1 (7.7) | 38.3 (11.1) | 37.7 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 14
  Male | 32 | 25 | 57
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 36 | 32 | 68
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 0 | 3
  White | 31 | 27 | 58
  More than one race | 2 | 6 | 8
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 38 | 33 | 71

OUTCOME MEASURES:

1. Primary Outcome: Recruitment
Description: Number of eligible participants who enrolled in the study
Time Frame: Assessed at baseline
Measure: Count of Participants; unit: Participants
Groups:
- Eligible Participants: Individuals who met all inclusion/exclusion criteria and were invited to participate in the study
Arm/Group | Eligible Participants
Number analyzed (Participants) | 92
Participants | 71

2. Primary Outcome: Retention
Description: Number of participants who complete all treatment sessions
Time Frame: Assessed at post-treatment (week 6)
Measure: Count of Participants; unit: Participants
Arm/Group | CBT-I | Sleep Hygiene
Number analyzed (Participants) | 38 | 33
Participants | 33 | 33

3. Primary Outcome: Drinking Quantity
Description: Assessed using Daily Drinking Questionnaire. Participants report the number of standard drinks consumed on each day of a typical week in the past month (on Monday, Tuesday, Wednesday, etc). Responses for each day are then summed to calculate a total "drinks per week" variable, where higher scores indicate more standard drinks.
Time Frame: Primary analyses will measure between-group change in at post (week 6) and follow-up (week 20). Mean values at each time point are presented below.
Population: Some participants lost to follow-up.
Measure: Mean (Standard Deviation); unit: drinks per week
Arm/Group | CBT-I | Sleep Hygiene
Number analyzed (Participants) | 38 | 33
drinks per week
  Baseline | 18.63 (15.76) | 17.94 (15.26)
  Post (week 6): number analyzed (Participants) | 31 | 26
  Post (week 6) | 15.29 (14.73) | 12.00 (9.84)
  Follow-up (week 20): number analyzed (Participants) | 33 | 30
  Follow-up (week 20) | 15.12 (21.96) | 15.73 (15.89)

4. Primary Outcome: Alcohol-related Consequences
Description: Assessed using the Brief Young Adult Alcohol Consequences Questionnaire, which asks participants to indicate (yes/no) which of 24 consequences they have experienced in the past month. Responses range from 0 to 24, with greater scores indicating more consequences.
Time Frame: as for outcome 3
Population: Some participants lost to follow-up.
Measure: Mean (Standard Deviation); unit: number of alcohol-related consequences
Arm/Group | CBT-I | Sleep Hygiene
Number analyzed (Participants) | 38 | 33
number of alcohol-related consequences
  Baseline | 7.92 (5.34) | 8.45 (6.49)
  Post (week 6): number analyzed (Participants) | 31 | 24
  Post (week 6) | 2.45 (3.25) | 4.46 (4.76)
  Follow-up (week 20): number analyzed (Participants) | 32 | 29
  Follow-up (week 20) | 3.31 (4.20) | 5.28 (4.35)

5. Primary Outcome: Insomnia Symptoms
Description: Assessed using Insomnia Severity Index (ISI). ISI scores from 0 to 28, with higher scores indicating more severe insomnia.
Time Frame: as for outcome 3
Population: Some participants lost to follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBT-I | Sleep Hygiene
Number analyzed (Participants) | 38 | 33
score on a scale
  Baseline | 17.29 (4.39) | 16.88 (4.15)
  Post (week 6): number analyzed (Participants) | 34 | 26
  Post (week 6) | 7.24 (4.83) | 12.27 (4.57)
  Follow-up (week 20): number analyzed (Participants) | 33 | 30
  Follow-up (week 20) | 6.97 (5.84) | 12.30 (5.14)

6. Primary Outcome: Sleep Quality
Description: On daily sleep diaries, participants reported sleep quality on a scale from 0 (very poor) to 4 (very good). Higher scores indicate better sleep quality.
Time Frame: as for outcome 3
Population: Some participants lost to follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBT-I | Sleep Hygiene
Number analyzed (Participants) | 38 | 33
score on a scale
  Baseline | 1.92 (0.60) | 1.73 (0.65)
  Post (week 6): number analyzed (Participants) | 32 | 24
  Post (week 6) | 2.49 (0.52) | 2.13 (0.87)
  Follow-up (week 20): number analyzed (Participants) | 26 | 23
  Follow-up (week 20) | 2.53 (0.63) | 2.14 (0.93)

7. Primary Outcome: Sleep Efficiency
Description: Daily sleep diaries were used to calculate the amount of time that participants spent sleeping out of all the time they spent in bed. Values from 0 to 100, with higher scores indicating better sleep efficiency. The treatment goal is 85%.
Time Frame: as for outcome 3
Population: Some participants lost to follow-up.
Measure: Mean (Standard Deviation); unit: percentage of time asleep
Arm/Group | CBT-I | Sleep Hygiene
Number analyzed (Participants) | 38 | 33
percentage of time asleep
  Baselin | 71.94 (11.84) | 68.82 (12.07)
  Post (week 6): number analyzed (Participants) | 32 | 24
  Post (week 6) | 87.89 (6.39) | 77.89 (8.84)
  Follow-up (week 20): number analyzed (Participants) | 26 | 23
  Follow-up (week 20) | 87.10 (9.57) | 79.90 (10.57)

8. Primary Outcome: Client Satisfaction
Description: Assessed using the 8-item Client Satisfaction Questionnaire. Participants rate their satisfaction with insomnia treatment on a scale from 1 (poor) to 4 (excellent). Scores were summed and then divided by the number of items to create a meaningful standardized score. Higher scores indicate greater satisfaction.
Time Frame: Mean score at post-treatment (week 6).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBT-I | Sleep Hygiene
Number analyzed (Participants) | 29 | 27
score on a scale | 3.59 (0.40) | 2.72 (0.57)

9. Secondary Outcome: Delay Discounting
Description: Assessed using the Monetary Choice Questionnaire (MCQ). Participants indicate if they would rather receive a smaller amount of money now or a greater amount of money in a specified amount of time (e.g., 100 days, 2 days). The MCQ is scored using a logarithmic subject-specific discount rate (k variable). K values typically fall between 0.0 and 0.5, with higher values indicating a preference for smaller, immediate rewards over larger, delayed reward ("delay discounting").
Time Frame: as for outcome 3
Population: Some participants were lost to follow-up.
Measure: Mean (Standard Deviation); unit: log (k)
Arm/Group | CBT-I | Sleep Hygiene
Number analyzed (Participants) | 36 | 33
log (k)
  Baseline | .028 (.062) | .022 (.046)
  Post (week 6): number analyzed (Participants) | 28 | 24
  Post (week 6) | .037 (.062) | .009 (.009)
  Follow-up (week 20): number analyzed (Participants) | 30 | 27
  Follow-up (week 20) | .033 (.062) | .011 (.014)

10. Secondary Outcome: Negative Affect
Description: Assessed using the Positive and Negative Affect Schedule. Participants indicate using a 1 (not at all) - 5 (extremely) scale to indicate to what extent they feel negative emotions. The final score is the sum of the ten negative emotions/feelings. Higher scores indicate more negative affect.
Time Frame: as for outcome 3
Population: Some participants lost to follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBT-I | Sleep Hygiene
Number analyzed (Participants) | 38 | 33
score on a scale
  Baseline | 16.82 (7.06) | 16.39 (6.82)
  Post (week 6): number analyzed (Participants) | 28 | 24
  Post (week 6) | 14.18 (5.19) | 18.29 (8.48)
  Follow-up (week 20): number analyzed (Participants) | 30 | 25
  Follow-up (week 20) | 15.77 (7.55) | 16.48 (5.67)

11. Secondary Outcome: Emotion Regulation
Description: Assessed using the Difficulties in Emotion Regulation Scale (DERS-16). Scores range from 0 to 64, with higher scores indicating more difficulties with emotion regulation.
Time Frame: as for outcome 3
Population: Some participants lost to follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBT-I | Sleep Hygiene
Number analyzed (Participants) | 38 | 33
score on a scale
  Baseline | 34.53 (13.22) | 32.85 (12.17)
  Post (week 6): number analyzed (Participants) | 28 | 24
  Post (week 6) | 27.14 (7.07) | 35.79 (12.54)
  Follow-up (week 20): number analyzed (Participants) | 30 | 25
  Follow-up (week 20) | 30.00 (11.49) | 34.88 (11.79)

12. Secondary Outcome: Alcohol Craving
Description: Assessed using the Penn Alcohol Craving Scale (PACS). Scores range from 0 to 30, with higher scores indicating more craving.
Time Frame: as for outcome 3
Population: Some participants lost to follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBT-I | Sleep Hygiene
Number analyzed (Participants) | 38 | 33
score on a scale
  Baseline | 9.29 (5.63) | 9.70 (6.82)
  Post (week 6): number analyzed (Participants) | 28 | 24
  Post (week 6) | 6.46 (5.91) | 7.62 (6.74)
  Follow-up (week 20): number analyzed (Participants) | 30 | 27
  Follow-up (week 20) | 7.30 (7.18) | 7.04 (5.96)

13. Secondary Outcome: Percentage of Days Using Alcohol to Help With Sleep
Description: Participants completed 2 weeks of sleep diaries assessing use of alcohol to help with sleep. Number of days reporting use of alcohol as a sleep aid was divided by the number of diaries completed to indicate the percentage of diary days they used alcohol as a sleep aid. Higher scores indicate more frequent use of alcohol as a sleep aid.
Time Frame: Primary analyses will measure between-group change at post (week 6) and follow-up (week 20). Mean values at each time point are presented below.
Population: Some participants lost to follow-up.
Measure: Mean (Standard Deviation); unit: % of diary days using alcohol for sleep
Arm/Group | CBT-I | Sleep Hygiene
Number analyzed (Participants) | 38 | 33
% of diary days using alcohol for sleep
  Baseline | 16.71 (27.86) | 6.73 (16.56)
  Post (week 6): number analyzed (Participants) | 32 | 24
  Post (week 6) | 3.22 (8.60) | 6.89 (22.94)
  Follow-up (week 20): number analyzed (Participants) | 26 | 23
  Follow-up (week 20) | 2.24 (4.88) | 9.12 (26.17)

14. Secondary Outcome: Percentage of Days Using Sleep Medication
Description: Participants completed 2 weeks of sleep diaries assessing use of sleep medication. Number of days reporting use of sleep medication was divided by the number of diaries completed to indicate the percentage of diary days they used a sleep medication. Higher scores indicate more frequent use of sleep medication.
Time Frame: as for outcome 13
Population: Some participants lost to follow-up.
Measure: Mean (Standard Deviation); unit: % of diary days using a sleep medication
Arm/Group | CBT-I | Sleep Hygiene
Number analyzed (Participants) | 38 | 33
% of diary days using a sleep medication
  Baseline | 30.92 (36.23) | 23.15 (35.49)
  Post (week 6): number analyzed (Participants) | 32 | 24
  Post (week 6) | 14.04 (30.71) | 28.44 (41.56)
  Follow-up (week 20): number analyzed (Participants) | 26 | 23
  Follow-up (week 20) | 11.55 (28.18) | 20.36 (38.35)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected through study completion, up to 22 weeks.
Arm/Group | CBT-I | Sleep Hygiene
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/33
Other Adverse Events (participants affected / at risk) | 1/38 | 0/33
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CBT-I (N=38) | Sleep Hygiene (N=33)
Unanticipated Problem Involving Risk (Psychiatric disorders) | 1 (1) | 0 (0) — Emotional distress in response to questionnaires

LIMITATIONS AND CAVEATS:
The COVID-19 pandemic changed the way people drink and required modifications to the protocol. Most treatment sessions were conducted via telehealth. As a result, all data were collected via self-report. Finally, data were collected from a relatively small, homogeneous sample of heavy-drinking Veterans. The control condition was not matched with CBT-I for time and content, so we cannot determine from this trial whether improvements are due to CBT-I or non-specific therapy effects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-29): https://cdn.clinicaltrials.gov/large-docs/88/NCT03804788/Prot_SAP_000.pdf